CLINICAL TRIAL: NCT00080457
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Safety and Efficacy Study of Sitaxsentan Sodium (Thelin™) Treatment With an Open-Label Bosentan Arm in Patients With Pulmonary Arterial Hypertension (PAH)
Brief Title: Safety and Efficacy Study of Sitaxentan Sodium (Thelin™) in Patients With Pulmonary Arterial Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Encysive Pharmaceuticals (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STRIDE 2
Record Dates: First submitted 2004-04-01; First posted 2004-04-05 (Estimated); Last update posted 2007-11-09 (Estimated); Status verified 2007-11

CONDITIONS: Pulmonary Hypertension
Keywords: Primary or secondary pulmonary arterial hypertension; Scleroderma; Connective tissue disease; Congenital heart defects; Lupus; Pulmonary Arterial Hypertension
MeSH Terms: conditions — Hypertension, Pulmonary; Scleroderma, Diffuse; Connective Tissue Diseases; Heart Defects, Congenital; Pulmonary Arterial Hypertension

INTERVENTIONS:
Drug: sitaxsentan sodium

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of Thelin™ (sitaxsentan sodium) compared to placebo (sugar pill) in the treatment of patients with pulmonary arterial hypertension (PAH).

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety and efficacy of Thelin™ (sitaxsentan sodium) as compared to placebo in the treatment of patients with PAH. A cohort of patients will be randomized to usual treatment with Tracleer® (bosentan) for observational comparisons of safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Have a current diagnosis of symptomatic PAH classified by one of the following:

  1. primary pulmonary hypertension (PPH) - also known as idiopathic pulmonary arterial hypertension (IPAH);
  2. PAH associated with connective tissue diseases;
  3. PAH associated with one of the following congenital heart defects:

     1. repaired ASD, VSD or PDA greater than one year post-operative
     2. un-repaired secundum ASD (with resting oxygen saturation greater than 88 percent in room air measured by oximeter)
* World Health Organization (WHO) functional class II, III, IV
* Greater than 12 and less than 75 years of age
* Women of childbearing potential must be using two forms of medically acceptable contraception (at least one barrier method)
* Have a cardiac catheterization within 6 months before study entry that shows the following values:

  1. mean pulmonary artery pressure (PAPm) greater than 25 mmHg (at rest),
  2. pulmonary capillary wedge pressure (PCWP) or left ventricular-end diastolic pressure less than 15 mmHg, and
  3. pulmonary vascular resistance (PVR) greater than 3 mmHg/L/min.

Exclusion Criteria:

* Portal hypertension or chronic liver disease
* ALT or AST levels greater than 1.5 times the upper limit of normal at the Screening Visit
* Contraindication to treatment with an endothelin receptor antagonist
* Recent history of abusing alcohol or illicit drugs
* Chronic renal insufficiency
* Pregnant or breastfeeding
* Atrial septostomy within 30 days before study entry
* Previous failure on bosentan because of safety concerns of the lack of clinical response

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 240
Dates: Start 2003-05; Study Completion 2005-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Encysive Pharmaceuticals, Houston, Texas, United States